CLINICAL TRIAL: NCT07059494
Title: A Feasibility Clinical Trial of Atezolizumab and Bevacizumab in Combination With Y^90 Radioembolization for Patients With Hepatocellular Carcinoma (HCC) for Liver Transplantation
Brief Title: Atezolizumab and Bevacizumab in Combination With Y^90 Radioembolization in HCC for Liver Transplant
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Principal Investigator, Parissa Tabrizian, Associate Professor of Surgery, Icahn School of Medicine at Mount Sinai
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY-24-01566; PRMC-24-146 (Other: PRMC)
Record Dates: First submitted 2025-06-17; First posted 2025-07-10 (Actual); Last update posted 2025-11-04 (Actual); Status verified 2025-11

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — atezolizumab; Bevacizumab

STUDY DESIGN:
Intervention Model Description: Feasibility study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cohort A: participants beyond Milan Criteria upon enrollment (Experimental): Atezolizumab and Bevacizumab in Combination with Y^90 Radioembolization
  Interventions: Drug: Atezolizumab; Drug: Bevacizumab; Radiation: Y^90 Radioembolization
- Cohort B: participants within Milan Criteria with AFP ≥ 400 ng/ml at enrollment. (Experimental): Atezolizumab and Bevacizumab in Combination with Y^90 Radioembolization
  Interventions: Drug: Atezolizumab; Drug: Bevacizumab; Radiation: Y^90 Radioembolization

INTERVENTIONS:
Drug: Atezolizumab — Atezolizumab is an immune checkpoint inhibitor. It is a monoclonal antibody that works by binding to the protein PD-L1 on the surface of some cancer cells, which keeps cancer cells from suppressing the immune system. It is indicated for usage in Non-Small Cell Lung Cancer (NSCLC), Small Cell Lung Cancer (SCLC), Hepatocellular Carcinoma (HCC), Melanoma, and Alveolar Soft Part Sarcoma (ASPS).
Drug: Bevacizumab — Bevacizumab is a vascular endothelial growth factor inhibitor indicated for the treatment of metastatic colorectal cancer, in combination with intravenous fluorouracil-based chemotherapy for first- or second-line treatment. It is also indicated for the treatment of metastatic colorectal cancer, in combination with fluoropyrimidine-irinotecan- or fluoropyrimidine-oxaliplatin-based chemotherapy for second-line treatment in participants who have progressed on a first-line bevacizumab product-containing regimen.
Radiation: Y^90 Radioembolization — Radioembolization is a minimally invasive procedure that combines embolization and radiation therapy to treat cancers in the liver. Tiny beads filled with a radioactive isotope are placed inside the blood vessels that supply a tumor. This blocks the supply of blood to the cancer cells and delivers a high dose of radiation to the tumor while sparing normal tissue. It can help extend the lives of participants with inoperable tumors and improve their quality of life.

SUMMARY:
A single institution, single arm, two-cohort feasibility trial to evaluate the combination of locoregional Y^90 therapy with systemic atezolizumab and bevacizumab, in participants presenting with hepatocellular carcinoma (HCC) 1) within Milan Criteria (MC) with AFP ≥ 400 ng/ml as a means of bridge therapy prior to transplant, 2) beyond the Milan Criteria (MC) (within USCF DS criteria and all comers), as a means of downstaging prior to liver transplantation.

DETAILED DESCRIPTION:
The researchers propose a single institution, single arm, two-cohort feasibility trial to evaluate the combination of locoregional Y^90 therapy with systemic atezolizumab and bevacizumab, in participants presenting with hepatocellular carcinoma (HCC) 1) within Milan Criteria (MC) with AFP ≥ 400 ng/ml as a means of bridge therapy prior to transplant, 2) beyond the Milan Criteria (MC) (within USCF DS criteria and all comers), as a means of downstaging prior to liver transplantation. Participants with macrovascular invasion and extrahepatic disease at diagnosis will be excluded from the study. Participants with AFP > 1000 ng/ml at diagnosis will be excluded.

ELIGIBILITY:
Inclusion Criteria:

* Signed Informed Consent Form
* Age ≥18 years at time of signing Informed Consent Form
* Ability to comply with the study protocol
* Newly diagnosed, biopsy-proven hepatocellular carcinoma (HCC) that is histologically or cytologically confirmed
* Availability of a representative tumor specimen that is suitable for determination of PD-L1 status via central testing. A formalin-fixed paraffin-embedded (FFPE) tumor specimen in a paraffin block (preferred) or 10-15 slides (15 slides preferred) slides containing unstained, freshly cut, serial sections should be submitted along with an associated pathology report prior to study enrollment. If archival tumor tissue is unavailable or is determined to be unsuitable for required testing, tumor tissue must be obtained from a biopsy performed at screening. Availability of a representative tumor specimen for exploratory biomarker research. Newly diagnosed, biopsy-proven hepatocellular carcinoma (HCC) either outside of the Milan Criteria (MC), or within the MC, with high risk disease as defined by alpha-fetoprotein (AFP) ≥400 ng/mL, and also fulfilling the criteria below.

  1. Within MC with AFP ≥ 400 ng/ml

     1. single lesion (≤5cm) or 3 lesions (≤3cm)
     2. Absence of vascular invasion or extra-hepatic disease based on cross-sectional imaging
     3. Child-Pugh Score of A/B7 (without ascites)
  2. UNOS-DS Protocol

     1. HCC exceeding UNOS T2 criteria but meeting one of the following:

        * Single lesion ≤ 8 cm
        * 2 or 3 lesions each ≤ 5 cm with the sum of the maximal tumor diameters ≤8 cm
        * or 5 lesions each ≤ 3 cm with the sum of the maximal tumor diameters ≤ 8 cm
     2. Absence of vascular invasion or extra-hepatic disease based on cross-sectional imaging
     3. Child-Pugh Score of A/B7 (without ascites)
  3. Beyond UNOS-DS Liver Only Protocol a. HCC exceeding UNOS-DS criteria by any of the following:

     * HCC tumor number
     * HCC tumor size
     * Total HCC tumor diameter b. Absence of vascular invasion or extra-hepatic disease based on cross-sectional imaging c. Child-Pugh Score of A/B7 (without ascites)
* Measurable disease, or non-measurable but evaluable disease, per RECIST v1.1 criteria
* Must meet institutional standards for proteinuria (Urinalysis (pH, specific gravity, glucose, protein, ketones, and blood); dipstick permitted
* Eligible for treatment with Y^90 and atezolizumab plus bevacizumab
* ECOG performance status of 0-1
* Life expectancy > 6 months
* Adequate hematologic and end-organ function, defined by the following laboratory test results, obtained within 14 days prior to initiation of study treatment:

  * ANC 1.5 ≥ 10^9/L (1500/µL) without granulocyte colony-stimulating factor support, with the following exception:
  * Participants with benign ethnic neutropenia (BEN): ANC < 1.3 x 10^9/L (1300/μL) BEN (also known as constitutional neutropenia) is an inherited cause of mild or moderate neutropenia that is not associated with any increased risk for infections or other clinical manifestations. BEN is referred to as ethnic neutropenia because of its increased prevalence in people of African descent and other specific ethnic groups.

    * Lymphocyte count ≥ 0.5 x 10^9/L (500/µL)
    * Platelet count ≥ 100 x 10^9/L (100,000/µL) without transfusion
    * Hemoglobin ≥ 90 g/L (9 g/dL)
  * Participants may be transfused to meet this criterion.

    * AST, ALT, and alkaline phosphatase (ALP) ≤ 2.5 upper limit of normal (ULN)
    * Serum bilirubin ≤ 1.5 x ULN with the following exception:
  * Participants with known Gilbert disease: serum bilirubin ≤ 3 x ULN

    * Serum creatinine ≤ 1.5 x ULN
    * Serum albumin ≥ 25 g/L (2.5 g/dL)
    * For participants not receiving therapeutic anticoagulation: INR or aPTT ≤ 1.5 x ULN
    * For participants receiving therapeutic anticoagulation: stable anticoagulant regimen
* Absent or controlled HIV, HCV, and HBV o Participants with a positive HIV test at screening are eligible provided they are stable on anti-retroviral therapy, have a CD4 count ≥ 200/μL, and have an undetectable viral load
* Negative serum pregnancy test within 14 days prior to the initiation of study treatment for participants of childbearing potential.
* Since adequate studies have not been performed in animals to determine whether Y^90 affects fertility in males or females has teratogenic potential or has other adverse effects on the fetus, this product should not be administered to pregnant or nursing women unless it is considered that the benefits to be gained outweigh the potential hazards. Ideally the use of this radioactive device in women of childbearing capability should be performed during the first few (approximately 10) days following the onset of menses.
* Agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive methods

Exclusion Criteria:

* AFP ≥ 1000 ng/ml
* Pathologically mixed tumors, vascular invasion or extra-hepatic disease based on cross-sectional imaging
* History of leptomeningeal disease
* Uncontrolled tumor-related pain

  o Participants requiring pain medication must be on a stable regimen at study entry.
* Severe pulmonary disease, uncontrolled pleural effusion, pericardial effusion, or ascites requiring recurrent drainage procedures (once monthly or more frequently) o Participants with indwelling catheters (e.g., PleurX®) are allowed
* Uncontrolled or symptomatic hypercalcemia (ionized calcium > 1.5 mmol/L, calcium > 12 mg/dL or corrected serum calcium > ULN)
* Active or history of autoimmune disease or immune deficiency, including, but not limited to, uncontrolled HIV, myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, antiphospholipid antibody syndrome, Wegener granulomatosis, Sjögren syndrome, Guillain-Barré syndrome, or multiple sclerosis (protocol lists a more comprehensive list of autoimmune diseases and immune deficiencies), with the following exceptions:

  * Participants with a history of autoimmune-related hypothyroidism who are on thyroid-replacement hormone are eligible for the study.
  * Participants with controlled Type 1 diabetes mellitus who are on an insulin regimen are eligible for the study.
  * Participants with eczema, psoriasis, lichen simplex chronicus, or vitiligo with dermatologic manifestations only (e.g., participants with psoriatic arthritis are excluded) are eligible for the study provided all of following conditions are met:

    * Rash must cover < 10 percent of body surface area
    * Disease is well controlled at baseline and requires only low-potency topical corticosteroids
    * There has been no occurrence of acute exacerbations of the underlying condition requiring psoralen plus ultraviolet A radiation, methotrexate, retinoids, biologic agents, oral calcineurin inhibitors, or high-potency or oral corticosteroids within the previous 12 months
* History of idiopathic pulmonary fibrosis, organizing pneumonia (e.g., bronchiolitis obliterans), drug-induced pneumonitis, or idiopathic pneumonitis, or evidence of active pneumonitis on screening chest computed tomography (CT) scan

  o History of radiation pneumonitis in the radiation field (fibrosis) is permitted.
* Active tuberculosis
* Significant cardiovascular disease (such as New York Heart Association Class II or greater cardiac disease, myocardial infarction, or cerebrovascular accident) within 12 months prior to initiation of study treatment, unstable arrhythmia, or unstable angina
* Major surgical procedure, other than for diagnosis or standard HCC care, within 4-6 weeks prior to initiation of study treatment, or during the study
* Core biopsy or other minor surgical procedure, excluding placement of a vascular access device, within 7 days prior to initiation of study treatment

  o Placement of a vascular access device should be at least 2 days prior to initiation of study treatment
* History of malignancy within 5 years prior to screening, with the exception of malignancies with a negligible risk of metastasis or death (e.g., 5-year overall survival (OS) rate > 90 percent), such as adequately treated carcinoma in situ of the cervix, non-melanoma skin carcinoma, localized prostate cancer, bladder cancer, carcinoma in situ, or Stage I uterine cancer
* Severe active infection within 4 weeks prior to initiation of study treatment, including, but not limited to, hospitalization for complications of infection, bacteremia, or severe pneumonia, active infection requiring IV antibiotics at the time of initiation of study treatment, or any active infection that could impact participant safety
* Treatment with therapeutic oral or IV antibiotics within 2 weeks prior to initiation of study treatment

  o Participants receiving prophylactic antibiotics (e.g., to prevent a urinary tract infection or chronic obstructive pulmonary disease exacerbation) are eligible for the study.
* Prior allogeneic stem cell, solid organ, or multi-organ transplantation
* Any other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding that contraindicates the use of an investigational drug, may affect the interpretation of the results, or may render the participant at high risk from treatment complications
* Treatment with a live, attenuated vaccine within 4 weeks prior to initiation of study treatment, or anticipation of need for such a vaccine during atezolizumab treatment or within 5 months after the final dose of atezolizumab
* Treatment with investigational therapy within 28 days prior to initiation of study treatment
* Prior treatment with CD137 agonists or immune checkpoint blockade therapies, including anti-CTLA-4, anti-PD-1, and anti-PD-L1 therapeutic antibodies
* Treatment with systemic immunostimulatory agents (including, but not limited to, interferon and interleukin 2 [IL-2]) within 4 weeks or 5 half-lives of the drug (whichever is longer) prior to initiation of study treatment
* Treatment with systemic immunosuppressive medication (including, but not limited to, corticosteroids, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-TNF-α agents) within 2 weeks prior to initiation of study treatment, or anticipation of need for systemic immunosuppressive medication during study treatment, with the following exceptions:

  * Participants who received acute, low-dose systemic immunosuppressant medication or a one-time pulse dose of systemic immunosuppressant medication (e.g., 48 hours of corticosteroids for a contrast allergy) are eligible for the study.
  * Participants who received mineralocorticoids (e.g., fludrocortisone), corticosteroids for chronic obstructive pulmonary disease (COPD) or asthma, or low-dose corticosteroids for orthostatic hypotension or adrenal insufficiency are eligible for the study.
* History of severe allergic anaphylactic reactions to chimeric or humanized antibodies or fusion proteins
* Known hypersensitivity to Chinese hamster ovary cell products or to any component of the atezolizumab formulation
* Known allergy or hypersensitivity to any component of the study therapy
* Prior locoregional or systemic therapy
* Pregnancy or breastfeeding, or intention of becoming pregnant during study treatment or within 6 months after the final dose of study treatment.
* Inadequately controlled hypertension (defined as systolic blood pressure > 150 mmHg and/or diastolic blood pressure > 100 mmHg)
* History of hypertensive crisis or hypertensive encephalopathy
* Significant vascular disease (e.g., aortic aneurysm requiring surgical repair or recent arterial thrombosis) within 6 months prior to randomization
* History of Grade ≥ 4 venous thromboembolism
* History or evidence upon physical or neurological examination of central nervous system involvement
* History of Grade ≥ 2 hemoptysis (defined as ≥ 2.5 mL of bright red blood per episode) within 1 month prior to screening
* History or evidence of inherited bleeding diathesis or significant coagulopathy at risk of bleeding (i.e., in the absence of therapeutic anticoagulation)
* History of abdominal fistula, GI perforation, intra-abdominal abscess, or active GI bleeding within 6 months prior to randomization
* Serious, non-healing wound, active ulcer, or untreated bone fracture
* Current or recent (< 10 days prior to initiation of study treatment) use of aspirin (> 325 mg/day), or clopidogrel (> 75 mg/day) Note: The use of full-dose oral or parenteral anticoagulants for therapeutic purpose is permitted as long as the INR and/or aPTT is within therapeutic limits (according to institution standards) within 7 days prior to initiation of study treatment and the participant has been on a stable dose of anticoagulants for ≥ 2 weeks prior to initiation of study treatment. Prophylactic use of anticoagulants is allowed. However, the use of direct oral anticoagulant therapies such as dabigatran (Pradaxa®) and rivaroxaban (Xarelto®) is not recommended due to bleeding risk.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-08-01 (Estimated); Study Completion 2028-08-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of Participants with Response to treatment | 9 months from first cycle of Y^90
  Cohort A Proportion of participants downstaging to within Milan Criteria as assessed by the rate of radiographic response via CT/MRI pre transplantation (efficacy window of assessment = 9 months from first cycle of Y^90)
  Cohort B Response rate to treatment in participants within MC with AFP ≥ 400 ng/ml defined by CT/MRI and a decrease in AFP ≥ 50 percent (efficacy window of assessment = 9 months from first cycle of Y^90)

SECONDARY OUTCOMES:
Adverse Events | 1 year
  All pre-transplant AEs and post-transplant related AEs will be summarized based on severity (based on CTCAE v5.0 grade), type of AE, and relationship to study treatment(s). A summary table of AEs will include the number and percentage of participants treated that experienced at least one: AE, SAE, Grade 3 or higher AE, Grade 4 or higher AE, treatment interruption, or dose reduction or treatment discontinuation. Rates of AEs will be calculated as the total number of AEs, SAEs, Grade 3 or higher AE, and Grade 4 or higher AEs per participant cycle on treatment. The analysis will be carried out in the SEAS population.
Pathological response | At time of transplant procedure
  Rate of pathological response at the time of transplantation (defined as >70 percent tumor necrosis at explant examination)
Disease progression | From time of treatment start to time of disease progression (at 1 year or upon occurrence of event, whichever comes first)
  Disease progression rate beyond baseline MC or post-downstage in participants beyond MC by CT/MRI (Cohort A).
  Disease progression is defined as per RECIST v1.1 and mRECIST staging criteria.
Recurrence-free survival (RFS) | From treatment Day 1 to post-transplant Year 1
  Assessment of efficacy of Y^90 in combination with atezolizumab and bevacizumab, pre- and post- transplant as defined Recurrence-free survival (RFS) rate at 1 year post LT, from time of study treatment start to first documented occurrence of intrahepatic or extra hepatic HCC using RECIST v1.1 and mRECIST criteria, or death from any cause, whichever occurs first.
Post-transplant recurrence rate | From Day 1 post-transplant to Year 1 post-transplant
  Assessment of efficacy of Y^90 in combination with atezolizumab and bevacizumab, pre- and post- transplant as defined by the Post-transplant recurrence rate at 1 year, from day 1 post-transplantation to first documented occurrence of intrahepatic or extra hepatic HCC using RECIST v1.1 and mRECIST criteria, or death, whichever occurs first.
Dropout rate from transplant waitlist | From treatment Day 1 to removal from transplant waiting list (i.e. disease progression, death) up to 3 years
  Assessment of efficacy of Y^90 in combination with atezolizumab and bevacizumab, pre- and post- transplant as defined by the Dropout rate from transplant waitlist
Rate of rejection of liver transplant | From Day 1 post-transplant to Year 1 post-transplant
  Assessment of efficacy of Y^90 in combination with atezolizumab and bevacizumab, pre- and post- transplant as defined by the Rate of rejection of liver transplant
Duration of response | from the first documentation of clinical/radiographical response, until death or progression, (at 1 year or upon occurrence of event) whichever comes first.
  The analysis of DOR will be performed on the ITT and PT populations. DOR is defined as time from the first documentation of clinical/radiographical response (per cohort definition of response) that is subsequently confirmed, to death or progression (as determined by the Investigator), whichever comes first. DOR will be censored at the date of last documentation of lack of death or disease progression for patients not known to have died or progressed at the time of data cutoff for analysis. DOR will be calculated only for the subset of patients with a response.
Time to the first response | Time of start of treatment to first documentation of cohort-defined clinical/radiographical response (at 1 year or upon occurrence of event, whichever comes first)
  Time to First response (TFR): Defined as time from the start of treatment to the first documentation of cohort-defined clinical/radiographical response that is subsequently confirmed. TFR will be calculated only for the subset of patients with a confirmed response. In this analysis, clinical/radiographical response (per cohort definition of response) will be the defining event while death without prior progression will be considered the competing event.

CONTACTS AND LOCATIONS:
Overall Officials: Parissa Tabrizian, MD, Principal Investigator — Mount Sinai Liver Cancer Program; Josep Llovet, MD, PhD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial, after deidentification.
Supporting Information: CSR
Time Frame: Immediately following publication. No end date.
Access Criteria: Investigators whose proposed use of the data has been approved by an independent review committee ('learned intermediary') identified for this purpose.
  To achieve aims in the approved proposal. Specify Other Mechanism Contact PI Parissa.Tabrizian@mountsinai.org